CLINICAL TRIAL: NCT06000163
Title: Normal Reference Values in Han Adults of Skin Thickness and Blood Flow by High-frequency Ultrasound: a Multicenter Study in China
Brief Title: Normal Reference Values in Han Adults of Skin Thickness and Blood Flow by High-frequency Ultrasound
Acronym: NOVAS-HFUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: NOVAS-HFUS-01
Record Dates: First submitted 2023-07-23; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteer; Skin
Keywords: skin thickness; dermal blood flow; high-frequency ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: high-frequency ultrasound — The volunteers will be given a high-frequency ultrasound examination of the skin, which is non-invasive, and skin thickness and blood flow parameters will be measured.

SUMMARY:
In recent years, high-frequency ultrasound has become a new non-invasive tool for the diagnosis of skin diseases, aesthetic medicine and preoperative and postoperative evaluation due to its higher resolution. The purpose of this multi-center Study is to establish the normal reference values of skin thickness and blood flow parameters by high-frequency ultrasound in Chinese Han adults, and to explore the influencing factors, so as to provide quantitative reference for the evaluation of facial skin aging degree and cosmetic treatment.

DETAILED DESCRIPTION:
The skin is the body's largest organ and acts as a protective, permeable barrier against pathogen invasion and against chemical and physical attacks. Long-term exposure to solar ultraviolet radiation is a major factor in exogenous skin aging. With the gradual improvement of living standards and the development of medical cosmetology technology, Chinese consumers have gradually increased their acceptance of cosmetology consumption. Facial skin, as one of the important indicators of "beauty", has obviously received the attention of cosmetic surgeons and dermatologists. Skin thickness is one of the important indicators of facial aging. However, different gender, different parts of the skin thickness is very different, especially the facial skin, the thickness of the epidermis, dermis is different, and the facial plastic surgery, injection treatment, photoelectric treatment has a close relationship. In addition, the dermis is rich in blood vessels, especially in its deep layers, which play an important role in the nutritional support of tissues and homeostasis of the internal environment. With the increase of age, the degree of dermal vascularization decreases, which is also one of the factors affecting skin aging. Therefore, in aesthetic medicine, more accurate quantitative evaluation of skin thickness and blood flow rather than simple subjective evaluation is very important.

Ultrasound is a non-invasive imaging technique widely used in clinic. In recent years, with the development of ultrasound technology, the frequency of ultrasonic probes has been increasing. Because of its higher resolution, high-frequency ultrasound can clearly display the layer and structure of the skin, and achieve accurate measurement of skin thickness and evaluation of dermal blood flow. High-frequency ultrasound has become a new non-invasive tool for the diagnosis of skin diseases, aesthetic medicine and preoperative and postoperative evaluation. The purpose of this multi-center Study is to establish the normal reference values of skin thickness and blood flow parameters by high-frequency ultrasound in Chinese Han adults, and to explore the influencing factors, so as to provide quantitative reference for the evaluation of facial skin aging degree and cosmetic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Han nationality;
2. Ages 18-79;
3. Normal blood pressure (139-90/89-60mmHg);
4. Body mass index < 30 kg/m2;
5. Blood routine, fasting blood glucose, blood lipid, liver and kidney function, electrocardiogram were normal;
6. No history of skin disease, connective tissue disease, cardiovascular disease, diabetes, severe liver and kidney dysfunction.
7. No history of drug use affecting cardiovascular system.

Exclusion Criteria:

1. People with skin diseases (such as eczema, psoriasis, scleroderma, etc.);
2. Any skin disease at the test site (such as dermatitis, acne, breakages, previous skin lesions, etc.);
3. chronic systemic diseases;
4. Use corticosteroid drugs or immunosuppressants;
5. Pregnant or lactating women;
6. People who have been exposed to ultraviolet radiation for a long time or have a history of sun exposure within 3 months;
7. The examined skin area has been previously treated with other methods;
8. Unable to cooperate with the inspector.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Chinese healthy Han adults
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Dermal thickness | 1 day
  Dermal thickness reflects the change in skin structure and can be used to assess skin aging.

SECONDARY OUTCOMES:
Blood flow velocity of dermal artery | 1 day
  Blood flow velocity of dermal artery reflects the hemodynamic changes of skin and can be used for early evaluation of skin aging.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine; Xinhua Ye, PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; WeiDong Ren, PHD, Principal Investigator — Shengjing Hospital; Xin Guan, PHD, Principal Investigator — Tianjin Chest Hospital; Hongning Yin, PHD, Principal Investigator — The Second Hospital of Hebei Medical University; Xiaoshan Zhang, PHD, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Yuhong Zhang, PHD, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University; Qingxiong Yue, PHD, Principal Investigator — Dalian Municipal Central Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-05-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT06000163/Prot_000.pdf
  • Informed Consent Form (2023-05-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT06000163/ICF_001.pdf